CLINICAL TRIAL: NCT04491487
Title: Effects of Pre-operative Speech-Language Pathology Counselling in Patients Undergoing to Total Laryngectomy: a Randomized Clinical Trial
Brief Title: Pre-operative Counselling in Laryngectomized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, LONGOBARDI YLENIA, researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3347
Record Dates: First submitted 2020-07-22; First posted 2020-07-29 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Total Laryngectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: pre-operative counselling
- Control group (No Intervention)

INTERVENTIONS:
Other: pre-operative counselling — pre-operative Speech-Language Pathology (SLP) counselling before Total Laryngectomy
  Arms: Experimental group

SUMMARY:
The investigators aim to verify the effects of pre-operative Speech-Language Pathology (SLP) counselling on patients undergoing total laryngectomy in terms of levels of distress, post-traumatic stress symptoms, anxious-depressive symptoms, acquisition and acceptance of the new voice.

This is a randomized controlled trial (RCT) of patients undergoing total laryngectomy and primary tracheoesophageal puncture. Patients will be randomized into two groups: an Experimental group that will receive a pre-operative SLP counselling session and a Control group that will not receive it. The investigators will administer a structured interview and three questionnaires: the Impact of Event Scale - Revised (IES-R), the Psychological Distress Inventory (PDI), the Hospital Anxiety and Depression Scale (HADS). The data will be collected between the 5th and 7th day after surgery (T0), 1-month (T1) and 3-months (T2) after being discharged from hospital.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years and over;
* patients waiting for TL and primary TEP;
* patients able and willing to provide written informed consent.

Exclusion Criteria:

* positive history for psychiatric or psychological disorders,
* neurological disorders,
* ineligibility for voice prosthesis rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Impact of Event Scale-revised | Between the fifth and seventh post-operative day (T0)
  presence of post-traumatic symptoms
Impact of Event Scale-revised | one month after being discharged from hospital (T1)
  presence of post-traumatic symptoms
Impact of Event Scale-revised | three months after being discharged from hospital (T2)
  presence of post-traumatic symptoms

SECONDARY OUTCOMES:
Psychological Distress Inventory | Between the fifth and seventh post-operative day (T0)
  psychological distress levels
Psychological Distress Inventory | one month after being discharged from hospital (T1)
  psychological distress levels
Psychological Distress Inventory | three months after being discharged from hospital (T2)
  psychological distress levels
Hospital Anxiety and Depression Scale | Between the fifth and seventh post-operative day (T0)
  anxiety and depression levels
Hospital Anxiety and Depression Scale | one month after being discharged from hospital (T1)
  anxiety and depression levels
Hospital Anxiety and Depression Scale | three months after being discharged from hospital (T2)
  anxiety and depression levels

CONTACTS AND LOCATIONS:
Overall Officials: Longobardi, Principal Investigator — Otolaryngology department
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No